CLINICAL TRIAL: NCT02179736
Title: A Post Market Evaluation After Treatment of Nasolabial Folds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05DF1312
Record Dates: First submitted 2014-06-19; First posted 2014-07-02 (Estimated); Last update posted 2022-08-25 (Actual); Status verified 2015-02

CONDITIONS: Nasolabial Folds
Keywords: Correction of moderate to severe nasolabial folds

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Active treatment (Experimental)
  Interventions: Device: Restylane

INTERVENTIONS:
Device: Restylane

SUMMARY:
This is an open, non-comparative study to evaluate effectiveness and safety of Restylane in correction of nasolabial folds up to 12 months after the initial treatment, and to evaluate the safety of repeat treatment of the nasolabial folds 12 months after the initial treatment.

ELIGIBILITY:
Inclusion Criteria

* 18 years or older
* Intent to undergo correction of both nasolabial folds
* WRSR 3-4
* Signed informed consent

Exclusion Criteria:

* Markedly indurate defects such as significant mid-face volume loss or prominent commissures.
* Active skin disease, inflammation or related conditions, such as infection, psoriasis and herpes zoster near or in the area to be treated.
* Subjects with known hypersensitivity to any ingredient of the study product or anaesthesia used in the study.
* Concomitant anticoagulant therapy and therapy with inhibitors of platelet aggregation, (e.g. non-steriodal anti-inflammatory drugs, acetylsalicylic acid, Omega 3 and Vitamin E) within 2 weeks prior to treatment, or a history of bleeding disorders.
* Concomitant treatment with chemotherapy, immunosuppressive agents, immunomodulatory therapy (e.g. monoclonal antibodies), systemic or topical (facial) corticosteroids. (Inhaled corticoids are allowed).
* Cancerous or pre-cancerous lesions in the treatment area.
* Subjects who have performed aesthetic facial surgery.
* Tissue augmenting therapy with non-permanent filler or neurotoxin below the lower orbital rim in the last 12 months.
* Facial laser treatment or chemical peeling below the lower orbital rim during the last 6 months.
* Permanent implant or filler, including fat-injections, placed in the area to be treated.
* Women who are pregnant or breast feeding or who are planning to become pregnant during the study period.
* Participation in any other clinical study within 30 days prior to inclusion.
* Any medical condition that in the opinion of the investigator would make the subject unsuitable for inclusion (e.g. a chronic, relapsing or hereditary disease that may affect the general condition or may require frequent medical treatment, psychiatric disorders or subjects not likely to comply to study procedures or to avoid other facial cosmetic treatments below the lower orbital rim).
* Subjects who are study site staff for this study, or close relatives (defined as parents, siblings, children or spouse) of the study site staff, as well as subjects who are employed by the sponsor company, or close relatives of employees at the sponsor company.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2014-07; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Effectiveness of study treatment in correction of nasolabial folds up to 12 months after a single treatment: | up to 12 months
  * Investigator evaluated wrinkle severity using wrinkle severity rating scale (WSRS)
  * Improvement in subject and investigator rated global aesthetic improvement (GAIS) compared to baseline.
  * Subject satisfaction

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Up to 12 months
  Safety of study treatment after single and repeat treatment of nasolabial folds will be assessed by:
  * Local tolerability (reported by subjects in a 14-day diary)
  * Adverse Events

CONTACTS AND LOCATIONS:
Locations (1):
- Plastic Surgery InstituteNo, No. 33 Badachu Road, Shijingshan District, Beijing Municipality, China